CLINICAL TRIAL: NCT04422509
Title: Lanadelumab for Treatment of COVID-19 Disease
Acronym: COVID_LAN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCN-AKF20.04
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — lanadelumab

STUDY DESIGN:
Intervention Model Description: controls will get standard of care and historical controls will be matched to the patients included
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lanadelumab (Experimental): 20 Patients will receive an intravenous dose of 300 mg lanadelumab on day 1, followed by a second dose of lanadelumab 300mg iv on day 4 (if needed).
  Interventions: Biological: lanadelumab
- controls (Other): 20 patients will received standard of care In additiona, for every index patient we will match one historical controls. Controls will be matched based on age, bodyweight and gender.
  Interventions: Other: regular care

INTERVENTIONS:
Biological: lanadelumab — single dose, or two doses administered iv
  Arms: lanadelumab
Other: regular care — no lanadelumab administration, treated according to regular care
  Arms: controls

SUMMARY:
So far little is very few drugs have demonstrated positive results for treatment of COVID19.

Recently the researchers have shown that the use of icatibant in COVID-19 results in a potent decrease in oxygen use. Yet the effect of the three dosages as according to the label dose was insufficient to maintain the clinical improvement in a small group of patients. The researchers argue that with the use of lanadelumab a more lasting effect can be reached due to its longer half life.

ELIGIBILITY:
Inclusion Criteria:

* Patient is SARS-COV2 positive (PCR)
* Without oxygen a saturation below 90%
* At least 3L/min oxygen dependent
* Patient is 16 years and older

Exclusion Criteria:

* Has previously participated in this study
* Acute myocardial or cerebral ischemic event at time of enrolment
* Receiving ACE or ARB inhibitor or comparable drugs that is specified as an intervention in this domain as a usual medication prior to this hospitalization will exclude a patient from receiving that agent
* A baseline alanine aminotransferase or an aspartate aminotransferase that is more than five times the upper limit of normal
* Patient is known hypersensitive to full human monoclonal antibodies
* Patient is pregnant or breast feeding

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
oxygen | 2 weeks
  oxygen use in L/min

SECONDARY OUTCOMES:
adverse events | 2 weeks
  adverse events after lanadelumab administration

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Amsterdam UMC, Amsterdam
  - Rijnstate hospital, Arnhem
  - Radboudumc, Nijmegen
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided
this has not yet been decided